CLINICAL TRIAL: NCT05985330
Title: Pilot Study of the Contribution of Fractional Exhaled Nitric Oxide as a Prognostic Marker of Response to Anti-PD-L1 Immunotherapy in Non-small Cell Lung Cancer
Acronym: FENOTYPE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GEORGES 2022
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients with metastatic non-small-cell lung cancer
  Interventions: Other: Measurement of FeNO

INTERVENTIONS:
Other: Measurement of FeNO — Before the first immunotherapy infusion and at the follow-up visit after the 4th course of immunotherapy

SUMMARY:
Based on the use of the patient's natural defences, immunotherapy mobilizes the immune system to recognize and destroy cancer cells, and it has revolutionized the treatment of lung cancer.

However, the effectiveness of immunotherapy varies from patient to patient. At present, we have no weak markers to predict with certainty the efficacy of immunotherapy treatment in a given individual.

Current scientific data identifies a number of molecules produced by the cancer cells and their environment which can be detected by various means (blood tests, breath analysis, etc.).

The aim of this study is to understand whether the amount of nitric oxide (NO) present in the breath is a more accurate predictor of response to immunotherapy.

Participation in this study involves breath testing (to measure FeNO (Fractional exhaled Nitric Oxide)) before receiving the first infusion of immunotherapy, and at the follow-up visit after the 4th course of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic NSCLC
* Patient not previously treated
* PD-L1 tumor expression > 50%, to be treated with immunotherapy alone after validation by a multidisciplinary consultation meeting.
* Patients over 18 years of age
* Patient having given his/her non-opposition
* Patient who speaks and reads French

Exclusion Criteria:

* Patients previously treated for NSCLC
* Patient with oncogene addiction or a first-line targetable rearrangement
* Patient not suitable for immunotherapy alone
* Patient having received corticosteroid treatment in the 15 days prior to FeNO.
* Patient on inhaled corticosteroid at time of inclusion.
* Blood eosinophilia > 500 /mm3
* Patient on 24-hour oxygen therapy
* Contraindication to immunotherapy
* Inability to perform FeNO measurement manoeuvres
* Pregnant, parturient or breast-feeding women
* Person under judicial protection (curatorship, guardianship)
* Person subject to limited judicial protection
* Adult unable to express their non-opposition
* Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic non-small-cell lung cancer requiring immunotherapy alone
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Response to immunotherapy by CT scan | after 4 courses of immunotherapy, an average of 9 weeks
  Evaluation according to RECIST criteria by comparing FeNO levels between patients responding and not responding to immunotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No